CLINICAL TRIAL: NCT02786667
Title: Non Motors Aspects in De Novo Parkinson's Disease: Clinical and Physiopathological Description; Dopamine Agonist Treatment Effects.
Brief Title: Non Motors Aspects in De Novo Parkinson's Disease
Acronym: Honeymoon
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-002855-33
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease; Apathy
MeSH Terms: conditions — Parkinson Disease; Lethargy | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): 6 months treatment with Rotigotine up to 8 mg per day with a titration period for one month
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): 6 months treatment with Placebo up to 8 mg per day with a titration period for one month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — 6 months treatment with Rotigotine up to 8 mg per day with a titration period for one month
  Other Names: Neupro
  Arms: Rotigotine
Drug: Placebo — 6 months treatment with Placebo up to 8 mg per day with a titration period for one month
  Arms: Placebo

SUMMARY:
Clinical description and pathophysiological study of recently diagnosed untreated patients with Parkinson's Disease.

Effect of a dopamine agonist (rotigotine) on apathy in de novo patients with Parkinson disease: A controlled, randomized, double blind study.

DETAILED DESCRIPTION:
This study aims to show the impact of a treatment with a D2/D3 receptor-specific dopamine agonist on the hypo-dopaminergic syndrome and quality of life of patients with de-novo Parkinson's disease.

The study consists of three parts:

1. The first part consists of a detailed clinical description of these patients, focusing on neuropsychological symptoms. The objective is to describe patients with and without apathy and hypo-dopaminergic syndrome.
2. From this population, a small number of patients with and without hypo-dopaminergic syndrome will be selected in order to compare serotoninergic and dopaminergic denervation by positron emission tomography (PET).
3. In patients with hypo-dopaminergic syndrome the motivational effects of a dopamine agonist will be tested in a randomized, double-blind, placebo-controlled study.

We hypothesize a significant improvement of apathy in the rotigotine group versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson disease without treatment for Parkinson disease
* Recent diagnosis (< 2 years)
* Without cognitive troubles

Exclusion Criteria:

* Patients with cognitive troubles
* Treated patients with L-Dopa or Dopamine agonists
* Other severe illness
* Pregnant or parturient woman

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of LARS (Lille Apathy Rating Scale) score in the rotigotine versus placebo group | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Castrioto, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No